CLINICAL TRIAL: NCT01354756
Title: Validation of Apnea LinkTM (ResMed Corporation, Poway, California) for Sleep Apnea Syndrome Screening in a Bariatric Population
Brief Title: Validation of Apnea LinkTM for Sleep Apnea Syndrome Screening in a Bariatric Population
Status: Terminated | Type: Observational
Why Stopped: device was stolen
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Chef de Clinique, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: AK/10-09-3921/52
Record Dates: First submitted 2011-05-06; First posted 2011-05-17 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Sleep Apnea Syndrome
Keywords: sleep apnea; polysomnography; obesity; bariatric surgery
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bariatric population: obese patients in whom a bariatric surgery is planified

SUMMARY:
Sleep apnea syndrome (OSA) frequently occurs in obese population undergoing bariatric surgery. There is a need for alternative screening tools for sleep apnea detection in the pre-operative period. The investigators would like to compare ApneaLink and complete polysomnography in this population.

DETAILED DESCRIPTION:
OSA can occur in up to 78% of patients undergoing bariatric surgery(1). Moderate to severe case will benefit from CPAP therapy, that can help avoiding post-operative complications(2).

In this population, the investigators propose complete attended in-hospital polysomnography (PSG)in patients with a clinical high probability of OSA.

According to obesity epidemics (3), waiting list for PSG in sleep labs is every day longer.

The investigators want to assess sensitivity and specificity of a new portable screening tool, ApneaLink, to detect OSA in a bariatric population.

Design:

monocentric and prospective study

Methods:

Patients:

- OSA suspicion based on :

* symptoms and signs (snoring, apneas , neck circumference >38 (women) or 43cm (men))
* BMI > 50
* BMI > 40, > 40 y
* BMI > 35, men, hypertension
* increased serum Bicarbonate
* Polyglobulia

Measurements

* Polysomnography in sleep lab with concommitant recording performed with Apnea LinkTM (nasal flow and oxymétry recording).
* between 2 weeks : recording performed with Apnea LinkTM (nasal flow and oxymétry recording)at home.

ELIGIBILITY:
Inclusion Criteria:

* obese patients
* > 18 years old
* in whom a bariatric surgery is planified and who have to undergo a polysomnography for OSA screening

Exclusion Criteria:

* pulmonary, neurologic, neuromuscular disease
* < 18 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese patients, > 18y old, in whom a bariatric surgery is planified and who have to undergo a polysomnography for OSA screening
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with correct diagnosis of OSA with ApneaLink. Therefore, we will compare apnea-hypopnea index measured with ApneaLink with apnea-hypopnea index measured during polysomnography. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, Principal Investigator — CHU St Pierre